CLINICAL TRIAL: NCT05162196
Title: Radiotherapy Combined With Niraparib and Toripalimab in Patients With Recurrent Small Cell Lung Cancer (CREATE): A Open-label, Single-arm, Phase II Study
Brief Title: The Efficacy and Safety of Radiotherapy Plus Niraparib and Toripalimab in Patients With Recurrent Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Conghua Xie,MD,PhD, Ph.D, Wuhan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREATE
Record Dates: First submitted 2021-12-04; First posted 2021-12-17 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Recurrent Small Cell Lung Cancer
Keywords: Radiotherapy; Toripalimab; Niraparib
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — toripalimab; niraparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT combined with Niraparib and Toripalimab (Experimental): Induction therapy (cyc1: D1-D28): Niraparib 200mg QD + SBRT 8Gy✖️3 QD, D4-D6 + Toripalimab 240mg iv drip D7
  Maintenance (cyc2+): Niraparib 200mg QD, D1-D21 + Toripalimab 240mg iv drip D1, until disease progression or intolerable toxicity
  Interventions: Radiation: SBRT; Drug: Toripalimab; Drug: Niraparib

INTERVENTIONS:
Radiation: SBRT — 24Gy/3F
Drug: Toripalimab — Toripalimab 240mg, ivgtt, d1, q3w.
Drug: Niraparib — 200mg qd

SUMMARY:
This is a prospective, multicenter, open-label study to observe the efficacy and safety of combination with radiotherapy, niraparib and toripalimab in patients With recurrent small cell lung cancer(SCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed small cell lung cancer.
2. Age ≥ 18 years.
3. Previously received 1-2 lines of treatment (including 1 systemic platinum-containing treatment), and responded to the first platinum-containing treatment (response is defined as CR, PR or SD).
4. At least 1 measurable target lesion based on RECIST 1.1.
5. Allow previous anti-PD-L1 antibody treatment, enrolled patients ≤ 30% of the total enrolled number.
6. Life expectancy ≥ 12 weeks.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status score 0-2.
8. Adequate hematologic function, hepatic function and renal function
9. Female who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must be willing to use an adequate method of contraception.
10. Male subjects of childbearing potential must agree to use an adequate method of contraception (failure rate < 1% per year) - Contraception, starting with the first dose of study therapy through 6 months after the last dose of study therapy.
11. . Toxic side effect to any previous chemotherapy has returned to ≤ CTCAE Grade 1 or baseline, or except sensory neuropathy or hair loss with stable symptoms ≤ CTCAE Grade 2.

Exclusion Criteria:

1. People who are known to be allergic to Niraparib or to active or inactive ingredients of drugs with similar chemical structure to Niraparib.
2. People who are known to be allergic to Toripalimab or to active or inactive ingredients of drugs with similar chemical structure to Toripalimab.
3. Symptomatic and uncontrolled cerebral or leptomeningeal metastasis. No imaging scan is required to confirm no brain metastases; subjects with spinal cord compression may be considered for inclusion if they have received targeted treatment and evidence of clinical stability of the disease for at least 28 days (patients with controlled CNS metastases must have received treatment such as radiotherapy or chemotherapy at least one month before entering the study; subjects should not develop new symptoms related to central nervous system lesions or symptoms indicating disease progression, and subjects either take stable doses of hormones or do not need to take hormones).
4. Chemotherapy or major surgery was performed within 3 weeks prior to the study or any surgical effect that has not been recovered after surgery.
5. Radiotherapy for target lesions within 4 weeks of initiating study drugs, or palliative radiotherapy for >20% bone marrow within 1 week prior to enrollment.
6. Patients with high risk of massive hemoptysis (such as uncured bronchiectasis, pulmonary tuberculosis).
7. Malignancies other than small cell lung cancer within 5 years prior to enrollment (except for radically treated cervical cancer in situ, basal cell carcinoma and superficial bladder tumor).
8. Patients with previously or currently diagnosed myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
9. Severe or uncontrolled conditions or diseases, including but not limited to:

   * Uncontrollable nausea and vomiting, inability to swallow study drugs, or any gastrointestinal disease that could affect drug absorption or metabolism.
   * Active virus infections such as human immunodeficiency virus (HIV) (positive HIV antibody), hepatitis B virus (HBV; positive HBsAg-positive status and HBV-DNA ≥10^3 copy number/mL or ≥500 IU/mL), and hepatitis C virus (HCV; positive anti-HCV antibody and/or positive HCV RNA in combination with clinical judgment).
   * Uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or mental disease impairing the participant's ability to give informed consent.
   * Known diagnosis of immunodeficiency (except for splenectomy) or other conditions that might predispose participants to a high risk of toxicity, as judged by the investigator.
10. Need to use any type of corticosteroids for systemic treatment within 14 days of study medication (>10mg/day prednisone) or other immunosuppressive drugs; in the absence of active autoimmune diseases, inhaled or topical steroids and Adrenal replacement dose (≤10mg/day prednisone); Allow patients to use topical, intraocular, intra-articular, intranasal and inhaled corticosteroids (small systemic absorption); allow physiological alternative doses of systemic corticosteroids (≤10mg/day prednisone); for prevention (such as contrast agents) Allergy) or short-term corticosteroid therapy for non-autoimmune diseases (such as delayed hypersensitivity caused by contact allergens) is allowed.
11. History of bleeding tendency and thrombosis:

    * Any bleeding events with CTCAE level 2 occurred within 3 months before screening, or with CTCAE level 3 and above within 6 months before screening
    * A history of gastrointestinal hemorrhage or a clear tendency of gastrointestinal hemorrhage within 6 months before screening. For example: esophageal varices with bleeding risk, local active ulcer lesions, or fecal occult blood + + or above
    * With active bleeding or coagulation abnormalities, bleeding tendency, or receiving thrombolytic or anticoagulation therapy
    * Subjects need anticoagulant therapy with warfarin or heparin
    * Subjects will require long-term antiplatelet therapy (e.g., aspirin, clopidogrel)
    * Thrombotic or embolic event within the past 6 months, e.g., cerebrovascular accident (including transient ischemic attack), and pulmonary embolism.
12. Serious cardiovascular history:

    * NYHA (New York Heart Association) grade 3 and 4 congestive heart failure
    * Unstable angina or newly diagnosed angina or myocardial infarction within 12 months before screening
    * Arrhythmias requiring therapeutic intervention (subjects taking β-blockers or digoxin may be enrolled)
    * ≥ CTCAE Grade 2 valvular heart disease
    * Poorly controlled hypertension (SBP > 150 mmHg or DBP > 100 mmHg).
13. Other laboratory abnormalities:

    * Hyponatremia (sodium <130 mmol/L); baseline serum potassium <3.5 mmol/L (potassium supplements can be used to restore serum potassium to above level before entering the study).
    * Abnormal thyroid function which cannot be maintained within the normal range with drugs.
14. Any previous or current disease, treatment or laboratory abnormality that may interfere with the results of the study, affect the subject's participation in the whole process of the research, or the researcher believes that the subject is not suitable for participating in this research; the subjects should not receive platelet or red cell transfusion within 4 weeks prior to the start of treatment with the study drug.
15. Subjects who are pregnant or breast-feeding or expect to become pregnant during the study treatment period.
16. Corrected QT interval (QTc)>450 milliseconds; if the subject has a prolonged QTc interval, but the investigator evaluates that the cause of the prolongation is a cardiac pacemaker (without other cardiac abnormalities), it is necessary to discuss with the investigator to determine whether the subject is suitable for inclusion in the study.
17. Previous treatment with any PARP inhibitors.
18. Previous treatment with any anti-PD-1 inhibitors.
19. Subjects are participating in other clinical studies or it is less than 1 month from the end of the previous clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
ORR (Objective response rate) | Approximately 2 years
  Objective response rate (ORR) evaluated by investigators and BIRC based on RECIST1.1

SECONDARY OUTCOMES:
DOR (Duration of Response) | Approximately 2 years
  Duration of response (DOR) evaluated by investigators and BIRC based on RECIST1.1
DCR (Disease of Response) | Approximately 2 years
  Disease control rate (DCR) evaluated by investigators and BIRC based on RECIST1.1
PFS (Progression Free Survival) | Approximately 2 years
  Progression free survival (PFS) evaluated by investigators according to the response evaluation criteria in solid tumors (RECIST 1.1)
PFS (Progression Free Survival) Rate | Approximately 1year
  PFS rates at 6-month（inestigators and BICR） and at 1-year
Overall suvival (OS) | Approximately 2 years
  Overall suvival (OS)
OS (Overall Survival) rate | Approximately 1 years
  OS rates at 1 years
Intrathoracic and extrathoracic recurrence rate | Approximately 2 years
The incidence of adverse events (AEs) as a measure of safety | Approximately 2 years
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered an investigational product. Safety and tolerance evaluated by incidence, severity and outcomes of AEs (according to NCI-CTCAE 5.0)

IPD SHARING:
Plan to Share IPD: No